CLINICAL TRIAL: NCT06217354
Title: Efficacy of Carbetocin at Elective Cesarean Section in Prevention of Postpartum Hemorrhage in Obese Versus Non-obese Women, A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Carbetocin in Prevention of Postpartum Hemorrhage in Obese Versus Non Obese Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Lecturer at Obstetrics and Gynecology department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Postpartum hemorrhage, Obesity
Record Dates: First submitted 2023-12-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Maternal; Post Partum Hemorrhage
MeSH Terms: conditions — Pregnancy in Obesity; Postpartum Hemorrhage | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Parturient with BMI ≥ 30 kg/m2. (Active Comparator): All patients will receive a bolus of carbetocin 100mcg IV over one minute after cord clamping. [PabalVR, Ferring AG, Baar, Switzerland]).
  Interventions: Drug: Carbetocin 100 Microgram/mL Solution for Injection
- Group B: Parturients with BMI < 30kg/m2 (control group) (Other): All patients will receive a bolus of carbetocin 100mcg IV over one minute after cord clamping. [Pabal, Ferring , Baar, Switzerland]).
  Interventions: Drug: Carbetocin 100 Microgram/mL Solution for Injection

INTERVENTIONS:
Drug: Carbetocin 100 Microgram/mL Solution for Injection — All patients will receive a bolus of carbetocin 100mcg IV over one minute after cord clamping. [PabalVR, Ferring AG, Baar, Switzerland]).then assess uterine contractility and postpartum bleeding measuring

SUMMARY:
Postpartum hemorrhage [PPH] can have serious consequences and is the leading cause of maternal mortality globally. Uterine contractility plays an important role in post-delivery uterine involution; impaired contractility can contribute to PPH. Should contractility be impaired among obese women, there would be implications for management. Therefore, the investigators sought to investigate whether obese women would also experience a need for more uterine agents during the management of an obstetric hemorrhage.

DETAILED DESCRIPTION:
The American College of Obstetricians and Gynecologists (ACOG) updated their definition of postpartum hemorrhage (PPH) to be "blood loss greater than or equal to 1000 ml or blood loss accompanied by signs or symptoms of hypovolemia" .

Recent clinical and translational studies have suggested a decrease in uterine contractility among obese and morbidly obese women as a primary cause of obstetric hemorrhage.

In the United States, the prevalence of maternal obesity has been steadily rising, with more than half of pregnant women classified as overweight or obese. A panel of obstetric experts has speculated that the rising prevalence of maternal obesity in developed countries may explain the increase in postpartum hemorrhage incidence.

Uterotonic drugs are recommended to reduce blood loss and the risk of postpartum hemorrhage (PPH) after Cesarean delivery.

There are several prophylactic uterotonic agents available for use, including oxytocin, oxytocin/ergometrine, and carbetocin. Carbetocin is a synthetic analog of oxytocin which provides a longer duration of action than oxytocin (half-life 85-100 min versus 3-4 min).

The investigators aim to investigate the impact of carbetocin on uterine contractility in obese versus non-obese pregnant women undergoing elective cesarean delivery following carbetocin 100 mcg bolus IV administration as a prophylaxis of postpartum hemorrhage in a randomized controlled trial. The incestigators hypothesize that increased volume of distribution reduces the bioavailability of carbetocin and may be an explanation for reduced efficacy. Also the investigators will examine uterine tone as a surrogate marker for the bioavailability of carbetocin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with a singleton pregnancy undergoing a Cesarean delivery after at least 37 completed weeks of gestation under regional anesthesia.
* Aged (18-39) years and with signed informed consent.

Exclusion Criteria:

* Emergency Cesarean Section due to fetal distress.
* Maternal comorbidities such as severe cardiovascular disorders, kidney or liver disorders, coagulopathies, as well as epilepsy.
* Uterine malformation.
* Fetal malformation.
* Known hypersensitivity to carbetocin or oxytocin.
* Uterine overdistention (as in polyhydramnios, twins, and fetal macrosomia)
* Injury of uterine vessels during CS.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Estimated Blood loss (ml) at cesarean section | 3 months
  Estimation of blood loss will be by assessing difference between pre -operative hemoglobin and a 24 hours after delivery hemoglobin and pre and 24h after delivery hematocrit according to the following formula: Estimated blood volume (pre-operative Hct-postoperative Hct)/pre-operative Hct.

SECONDARY OUTCOMES:
Uterine contractility and the need for more doses of carbetocin | 3 months
  Uterine contractility, the proportion of women receiving additional uterotonics after administration of single dose of carbetocin, transfusion of blood products and use of non-drug measures to treat PPH.
Estimated Blood loss by weighing gauze towel | 3 months
  weighing gauze towels (grams)pre and postoperative. Using suction when amniotic fluid membranes rupture up to delivery of the placenta. Gauze towels will be used exclusively to mop up the blood until closure of the abdomen

CONTACTS AND LOCATIONS:
Locations (1):
- Shaimaa El Shemy, Giza, Cairo Governorate, Egypt